CLINICAL TRIAL: NCT05202821
Title: Clinical Evaluation of the Efficacy of SPR-G (Surface Pre-reacted Glass Ionomer) Barrier Coat Versus Fluoride Varnish Versus the MI Paste (CPP-ACP) in the Treatment of Early White Spot Lesions in Pediatric Patients
Brief Title: Clinical Evaluation of the Efficacy of SPR-G Barrier Coat Versus Fluoride Varnish Versus MI Paste in the Treatment of Early White Spot Lesions in Pediatric Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Alsagheer, Master's Candidate, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 18-7M
Record Dates: First submitted 2021-03-01; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: White Spot Lesions [Initial Caries] on Smooth Surface of Tooth
Keywords: White spot lesions; Fluoride varnish; MI paste (CPP_ACP); SPRG- Barrier coat
MeSH Terms: interventions — PRG Barrier Coat; cavity shield; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- group of 20 participants receiving fluoride varnish (Active Comparator): *Group (I): patients will receive Fluoride varnish ttt.
  Interventions: Drug: Fluoride varnish
- group of 20 participants receiving PR-G Barrier coat (Experimental): *Group (II): patients will receive PR-G Barrier coat
  Interventions: Drug: PRG Barrier Coat
- group of 20 participants receiving MI Paste (CPP-ACP) (Active Comparator): *Group (III): Patients will receive MI Paste (CPP-ACP)
  Interventions: Drug: MI paste

INTERVENTIONS:
Drug: PRG Barrier Coat — 3 arm randomized single blind clinical trial comparing 3 groups. first group will be receiving fluoride varnish, second group will be receiving PRG Barrier Coat and the third group will be receiving MI paste
  Other Names: SPRG Barrier Coat
  Arms: group of 20 participants receiving PR-G Barrier coat
Drug: Fluoride varnish — First group will be receiving Fluoride varnish every 3 months
  Other Names: Cavity Shield
  Arms: group of 20 participants receiving fluoride varnish
Drug: MI paste — Third group will be receiving MI paste
  Other Names: RECALDENT™; (CPP-ACP)
  Arms: group of 20 participants receiving MI Paste (CPP-ACP)

SUMMARY:
In-Vivo randomized clinical trial to compare between the clinical performance of fluoride varnish versus MI paste (CPP_ACP) and the PRG- Barrier coat material concerning enamel remineralization, arrest of active early lesions, resolution of inactive incipient lesions and patient satisfaction and motivation with a 9-months follow up using a high resolution Nikon camera with Canon 700D body. Canon EF 100mm f2.8 USM Macro Lens and Nissin MF18 ring flash Canon fit for better illumination. Also, A set of retractors and A set child occlusal mirrors with A contraster for assessment of the remineralization progress of the white spot lesion.

DETAILED DESCRIPTION:
A total of sixty (60) patients with early white spot lesions will be randomly selected to share in this study from the out-patient clinic of pedodontics and orthodontic department, Faculty of dentistry, Ain Shams University.

An informed consent will be signed by the patients and parents before their enrollment in the current study in which the aim of the study, the methodology and possible complications will be clearly described. This research will be reviewed by the research ethics committee, Faculty of dentistry, Ain Shams University. This In-vivo study will aim to evaluate the effectiveness of the SPR-G filler material sealants when compared to the fluoride varnish and the MI paste.

Precise medical, dental and family history will be taken from all patients through a direct interview and diagnostic sheet.

Teeth will be polished using a polishing brush and paste, and dried thoroughly before being examined.

Clinical examination will be done using a dental mirror and aided by the tactile detection of a dental explorer under LED illumination to make sure that the patients fulfill the inclusion criteria, followed by radiographic examination. All examination and follow up procedures will be done by the same operator to ensure standardization.

Patient's Grouping:

Selected patients will be randomly divided into three groups:

* Group (I): patients will receive Fluoride varnish ttt.
* Group (II): patients will receive PR-G Barrier coat
* Group (III): Patients will receive MI Paste (CPP-ACP)

Patients who fail to show up at the follow up examinations will be automatically excluded from the study. Patients who are no longer willing to continue in the study will have the right to quit at any time.

Patient information will be gathered and stored in the patient examination chart of the outpatient clinic, Department of Pediatric Dentistry, faculty of Dentistry, Ain Shams University. All information will be kept as a hard copy and as an electronic one as well. Patient information will be guarded as confidential information that should never be revealed at all times. This file will remain with the investigator during the study.

Outcome measurement:

9 months' in vivo evaluation of functional & biological aspects of the three modalities regarding retention, stability, oral hygiene and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-16 years old
* Patient is healthy and medically free.
* Moderate to high level of patient cooperation
* Compliance of the primary caregiver
* Moderate to high caries risk
* Completed or in transitional fixed orthodontic treatment
* At least 1 wsl should be present

Exclusion Criteria:

* Poor oral hygiene
* Deeply Cavitated white spot lesions
* Medically Compromised patients.
* Extremely Uncooperative patient or primary caregiver
* Generalized white spot lesions in the mouth

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the size of the white spot lesions using photographic assessment | 9 months
  participants are divided into 3 groups. Each group receiving a different management approach to find out the most effective drug in reducing the size of white spot lesions. Photos are taken pre-operatively. 1 month, 3 months and 9 months

SECONDARY OUTCOMES:
Remineralization of the enamel surface | 9 months
  Using photographic assessment with the aid of a software to asses the change in the height and width (i.e surface area) of the white spot lesion

OTHER OUTCOMES:
Patient satisfaction and motivation towards treatment using a questionnaire at the end of the treatment | 9 months
  Closed ended questions with strongly agree rated with 5, agree rated 4, neutral rated 3, disagree rated 2 and strongly disagree rated 1. Higher values will denote positive results lower values indicating negative results

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abd El Aziz, Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Al Waili, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 9 months